CLINICAL TRIAL: NCT04098549
Title: The Effect of Rapid and Slow Glucose Fall on the Subsequent Glucose Production in People With Type 1 Diabetes
Acronym: RaSlo-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-19034585
Record Dates: First submitted 2019-09-11; First posted 2019-09-23 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Type 1 Diabetes; Blood Glucose, Low; Glucose Metabolism Disorders
Keywords: Type 1 Diabetes; Glucose Metabolism; Hypoglycemia; Glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Hypoglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid-Slow (Experimental): This arm will begin with intervention "rapid" (rapid rate of fall in plasma glucose) for the first study visit and proceed to intervention "slow" (slow rate of fall in plasma glucose) for the second study visit.
  Interventions: Other: Rapid lowering of plasma glucose; Other: Slow lowering of plasma glucose
- Slow-Rapid (Experimental): This arm will begin with intervention "slow" (slow rate of fall in plasma glucose) for the first study visit and proceed to intervention "rapid" (rapid rate of fall in plasma glucose) for the second study visit.
  Interventions: Other: Rapid lowering of plasma glucose; Other: Slow lowering of plasma glucose

INTERVENTIONS:
Other: Rapid lowering of plasma glucose — Rapid lowering of plasma glucose using hypoglycemic clamp technique
Other: Slow lowering of plasma glucose — Slow lowering of plasma glucose using hypoglycemic clamp technique

SUMMARY:
In the effort of better understanding the glucose control in people with type 1 diabetes, in-depth insight into the physiology of hepatic glucose production and its influencing factors is essential. Previously, a number of potential influencing factors of hepatic glucose production have been investigated, including insulin-on-board, low carbohydrate diet, preceding ethanol intake, exercise and multiple stimulations of hepatic glucose production. Previous post-hoc analysis of dual-hormone closed-loop systems has indicated that the rate of fall in blood glucose influences the following stimulation of hepatic glucose response. However, the rate of fall in blood glucose is highly related to insulin levels, which may explain those findings. Thus, in this study the investigators want to examine whether the different rates of fall in blood glucose with similar insulin levels on board affect the hepatic glucose response in individuals with type 1 diabetes. In the study, which will be conducted at Steno Diabetes Center Copenhagen, participants will complete two study visits. On each visit, a hypoglycemic clamp technique will be used to lower the blood glucose levels of the participants (using either a rapid or slow decline rate), whereupon hepatic glucose production will be stimulated using low-dose glucagon. The study days are divided into four phases: 1) preparation phase, 2) hyperinsulinemic euglycemic phase (stabilization of blood glucose), 3) hyperinsulinemic hypoglycemic phase (rapid or slow decline in blood glucose) and 4) post-glucagon administration phase. This design will allow the investigators to examine whether differences in hepatic glucose response exist depending on preceding rate of fall in blood glucose. We hypothesize that the rate of fall in blood glucose does not affect the hepatic glucose production.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Duration of Type 1 Diabetes ≥ 3 years
* Insulin pump use > 6 months

Exclusion Criteria:

* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start
* Allergy or intolerance to lactose or GlucaGen (Novo Nordisk, Bagsværd, DK)
* Use of medications that are known to cause QT interval prolongation
* Females who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods
* Females who have different basal insulin pattern depending on their menstrual cycle
* Inability to understand the individual information and to give informed consent
* Current participation in another clinical trial that, in the judgment of the principle investigator, will compromise the results of the study or the safety of the subject
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the individual unsuitable for study participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Positive incremental area under the glucose curve (PI-AUC) (using the plasma glucose concentration before glucagon administration as basal level) | from 0-120 minutes after glucagon administration

SECONDARY OUTCOMES:
Total area under the glucose curve (AUC) | from 0-120 minutes after glucagon administration
Peak plasma glucose | from 0-120 minutes after glucagon administration
Incremental plasma glucose peak | from 0-120 minutes after glucagon administration
Time-to-peak plasma glucose | from 0-120 minutes after glucagon administration
Plasma glucose level | 120 minutes after glucagon administration
Duration of plasma glucose above 4.0 mmol/l | from 0-120 minutes after glucagon administration
Duration of plasma glucose above baseline | from 0-120 minutes after glucagon administration
Number of subjects who, after reaching a plasma glucose value > 3.9 mmol/l following glucagon administration, maintain a plasma glucose level in the range of 3.9-10 mmol/l | throughout phase 4 (until 120 minutes after glucagon administration)
Number of subjects who, after reaching a PG > 3.9 mmol/l following glucagon administration, maintain a plasma glucose level in the range of 3.9-7.8 mmol/l | throughout phase 4 (until 120 minutes after glucagon administration)
Time from glucagon administration to reaching a plasma glucose level > 3,9 mmol/l | from 0-120 minutes after glucagon administration
Duration of a plasma glucose level in the range of 3.9-10 mmol/l | from 0-120 minutes after glucagon administration
Duration of a plasma glucose level in the range of 3.9-7.8 mmol/l | from 0-120 minutes after glucagon administration
Change in insulin levels (measured as area under the curve) | 0-120 minutes after glucagon administration
Change in insulin levels (measured as peak change) | from baseline to 120 minutes after glucagon administration
Change in glucagon levels (measured as area under the curve) | 0-120 minutes after glucagon administration
Change in glucagon levels (measured as peak change) | 0-120 minutes after glucagon administration
Average changes in Edinburgh Hypoglycemia Scale | measured at baseline, 5 minutes prior to the end of phase 2, 5 minutes prior to the end of phase 3 and 30 and 115 minutes after glucagon administration
Average change in visual analogue scale score for nausea, headache, stomach ache and palpitations | measured at baseline, 5 minutes prior to the end of phase 2, 5 minutes prior to the end of phase 3 and 30 and 115 minutes after glucagon administration
Number of subjects experiencing vomiting | from 0-120 minutes after glucagon administration

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol